CLINICAL TRIAL: NCT05322941
Title: A Multicenter, Double-blind, Placebo-controlled, Randomized, Parallel-group, Phase 2b Study in Treatment-seeking Patients With Cannabis Use Disorder to Assess the Efficacy, Safety, and Tolerability of AEF0117 in Reducing Cannabis Use
Brief Title: Effect of AEF0117 on Treatment-seeking Patients With Cannabis Use Disorder (CUD)
Acronym: SICA2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aelis Farma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AEF0117-202
Record Dates: First submitted 2022-03-24; First posted 2022-04-12 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Marijuana Abuse
Keywords: AEF0117; Cannabis-related Use Disorder; Cannabis subjective effects; Cannabis self-administration cannabis-induced analgesia; Cannabis-related cognitive disorder
MeSH Terms: conditions — Marijuana Abuse

STUDY DESIGN:
Intervention Model Description: Up to 330 eligible male or female subjects will be randomized into 1 of 4 treatment groups. The number of females to be enrolled will be limited to ensure that a maximum of 80 female subjects are assigned to active treatment (i.e., to 1 of the AEF0117 treatment groups).
  Subjects will be randomized to 1 of 4 treatment groups:
  * AEF0117 1.0 mg once daily (QD) (90 subjects)
  * AEF0117 0.3 mg QD (90 subjects)
  * AEF0117 0.1 mg QD (60 subjects)
  * Placebo (90 subjects)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AEF0117 (Experimental): The current study tests 3 doses of AEF0117 (1.0, 0.3, and 0.1 mg).AEF0117 capsules ; dose range 0.1 to 1.0mg by mouth, once a day for 12 weeks.
  Interventions: Drug: AEF0117
- Placebo (Placebo Comparator): corn oil capsules once a day for 12 weeks.
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: AEF0117 — AEF0117 (1.0, 0.3, and 0.1 mg) capsules
  Other Names: 3ß-(4-methoxybenzyloxy)pregn-5-en-20-one
  Arms: AEF0117
Drug: Placebo oral capsule — Corn oil capsule manufactured to mimic AEF0117 capsule
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
Cannabis use is increasing and will only further escalate with legalization of recreational and medical cannabis use in western countries , with a prevalence greater than 30 % in the US and most European countries for individuals between 16 and 24 years of age. Approximately 9 % of those who use cannabis will become addicted. The number goes up to about 1 in 6 among those who start using cannabis as teenagers and to 25 to 50 % among those who smoke cannabis daily. The consequences of cannabis abuse in the most prone population (14-25 years of age) are extremely serious, and may include addiction, altered brain development, poorer educational outcomes, cognitive impairment, lower income, greater welfare dependence, unemployment and lower relationship and life satisfaction. There are no available pharmacological treatments of cannabis use disorder (CUD). Thus, the development of safe and effective medications for the treatment of CUD is an urgent public health priority.

The preclinical efficacy and available ADMET (Administration, Distribution, Metabolism, Elimination and Toxicology) in animal and human data suggest that AEF0117, an investigational new study drug, could constitute a very efficacious and safe treatment for cannabis abuse disorders. The purpose of this research is to study how AEF0117 influences the subjective effects of cannabis in subjects with CUD. AEF0117 acts in the same parts of the brain as THC (tetrahydrocannabinol), the active ingredient of marijuana, and may temporarily alter some of cannabis's effects.

The safety and tolerability of AE0117 has been demonstrated in the clinical studies conducted to date. This study will provide additional data on the efficacy of AEF0117 on treatment-seeking subjects with moderate to severe CUD.

This is a phase 2b, randomized, double-blind, placebo-controlled, 4-arm, parallel-group, prospective, multicenter study. The overall purpose of this study is to assess the efficacy and safety of AEF0117 in subjects with moderate to severe CUD who are treatment-seeking. The primary objective of this study is to demonstrate that AEF0117 induces a greater proportion of RESPONDERS (i.e., subjects with a RESPONSE of ≤1 day of cannabis use per week) compared to placebo in treatment-seeking subjects with moderate to severe CUD, according to DSM-5 criteria.The secondary objectives are to investigate the proportion of subjects that reach various levels of reduction and how this influences their quality of life, and to evaluate the safety and tolerability of AEF0117. And the exploratory objectives of this study are to further evaluate the effect of AEF0117 on pattern of cannabis use and change in various signs and symptoms, and in addition to assess effects during the grace period and the entire treatment period.

DETAILED DESCRIPTION:
Cannabis use is increasing and will only further escalate with legalization of recreational and medical cannabis use in western countries , with a prevalence greater than 30 % in the US and most European countries for individuals between 16 and 24 years of age. Approximately 9 % of those who use cannabis will become addicted. The number goes up to about 1 in 6 among those who start using cannabis as teenagers and to 25 to 50 % among those who smoke cannabis daily. The consequences of cannabis abuse in the most prone population (14-25 years of age) are extremely serious, and may include addiction, altered brain development, poorer educational outcomes, cognitive impairment, lower income, greater welfare dependence, unemployment and lower relationship and life satisfaction. There are no available pharmacological treatments of cannabis use disorder (CUD). Thus, the development of safe and effective medications for the treatment of CUD is an urgent public health priority.

The preclinical efficacy and available ADMET (Administration, Distribution, Metabolism, Elimination and Toxicology) in animal and human data suggest that AEF0117, an investigational new study drug, could constitute a very efficacious and safe treatment for cannabis abuse disorders. The purpose of this research is to study how AEF0117 influences the subjective effects of cannabis in subjects with CUD. AEF0117 acts in the same parts of the brain as THC (tetrahydrocannabinol), the active ingredient of marijuana, and may temporarily alter some of cannabis's effects.

The safety and tolerability of AE0117 has been demonstrated in the clinical studies conducted to date. This study will provide additional data on the efficacy of AEF0117 on treatment-seeking subjects with moderate to severe CUD.

This will be a phase 2b, randomized, double-blind, placebo-controlled, 4-arm, parallel-group, prospective, multicenter study. The overall purpose of this study is to assess the efficacy and safety of AEF0117 in subjects with moderate to severe CUD who are treatment-seeking. The overall purpose of this study is to assess the efficacy and safety of AEF0117 in subjects with moderate to severe CUD who are treatment-seeking.

Up to 330 eligible male or female subjects will be randomized into 1 of 4 treatment groups. Due to the difference in prevalence of CUD between males and females, the number of females enrolled is anticipated to be less than 1/3 of all subjects. Moreover, the number of female subjects to be enrolled will be limited via stratification ensuring that a maximum 80 females will be assigned to active treatment (i.e., to 1 of the AEF0117 treatment groups), considering the development stage of the compound.

Subjects will be randomized to 1 of 4 treatment groups:

* AEF0117 1.0 mg once daily (QD) (90 subjects)
* AEF0117 0.3 mg QD (90 subjects)
* AEF0117 0.1 mg QD (60 subjects)
* Placebo QD (90 subjects)

The primary objective of this study is to demonstrate that AEF0117 induces a greater proportion of RESPONDERS (i.e., subjects with a RESPONSE of ≤1 day of cannabis use per week) compared to placebo in treatment-seeking subjects with moderate to severe CUD, according to DSM-5 criteria.

The secondary objectives are to investigate the proportion of subjects that reach various levels of reduction and how this influences their quality of life, and to evaluate the safety and tolerability of AEF0117.

* Assess if AEF0117 increases the proportion of subjects that reach complete abstinence (0 cannabis use).
* Assess if AEF0117 increases the proportion of subjects that have a modest level of cannabis use (≤2 days per week).
* Assess if AEF0117 increases the proportion of subjects that report no CUD symptoms according to DSM-5 except for craving (modified early remission, which is defined by the same criteria of the DSM-5 but without the required minimal time duration of the remission).
* Assess if AEF0117 decreases the percentage of days of cannabis use.
* Assess if AEF0117 improves the quality of life as measured by the Patient-Reported Outcomes Measurement Information System-29 (PROMIS-29) adult profile.
* Assess if AEF0117 introduce a change in pattern of cannabis use over the day.
* Assess the safety and tolerability of AEF0117.

The exploratory objectives of this study are to further evaluate the effect of AEF0117 on pattern of cannabis use and change in various signs and symptoms, and in addition to assess effects during the grace period and the entire treatment period.

The study consists of a screening period, a double-blind treatment period which includes a grace period and a treatment ascertainment period, and a follow-up period. The study will be conducted on an outpatient basis at the sites with a total of 27 visits per subject after screening for eligibility. During the 12-week treatment period, 25 visits will be performed: 1 weekly visit will include most of the scheduled assessments (13 full visits), while the second weekly visit will only include few assessments (12 short visits).Under certain circumstances, a short visit may be converted to a remote visit if it does not pose a risk to the safety of the subject as judged by the investigator.

During the 4-week follow-up period, 2 visits approximately 14 days apart will take place.

The double-blind randomized treatment period will consist of 2 periods: a 4-week grace period and an 8-week treatment ascertainment period. During both periods, subjects will attend standardized medical management sessions once a week with trained professionals (i.e., 12 visits in total).

During the grace period (Day 1 to Day 28), cannabis use will not be a criterion for characterization of non-responding subjects. This period will allow AEF0117 to reach plasma steady state and allow for behavioral changes. During the treatment ascertainment period (Day 29 to Day 84), any cannabis use will be taken into consideration to assign subjects as responders and non-responders.

All study visits will be conducted on an outpatient basis at the sites. Screening visit(s), weekly full visits during the grace period and treatment ascertainment period (13 visits) and visits every second week during follow up (2 visits) include extended assessments. In addition, 1 short visit per week is scheduled during the grace period and treatment ascertainment period (12 visits), including a few assessments (the second of the twice weekly visits).

Efficacy will be assessed using different observer-rated and self-reported scales.

Self-reported cannabis use will be monitored daily, prospectively by an Ecological Momentary Assessment (EMA) using a smartphone-based application and retrospectively by using the TLFB procedure.

The documentation of self-reported cannabis use will be based primarily on the EMA data and, in the case of missing data, on the TLFB data. In the case of a discrepancy, the more conservative data will be used (i.e., presence of an episode of use).

Adverse events will be monitored by research staff and medical observations and spontaneous reporting throughout the study. The grading system of adverse events used in this study will be the grading system proposed by Sibille M., et. al. Specifications on the grading system for clinical observations and ECG parameters will be based on the publication by Sibille M, Patat A, et al. Vital signs and laboratory parameters will be based on the FDA vaccine guidance (The Biologics Blood Vaccines Guidance Compliance, FDA).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects between 18 and 65 years old, both inclusive.
2. Subjects must meet DSM-5 criteria for moderate to severe CUD as assessed by the standard MINI-5.
3. Subjects must be treatment-seeking and have a mean cannabis use of ≥5 days per week within the last 4 weeks at the screening and baseline visit of the study. Mean cannabis use is assessed by the TLFB and a positive urine concentration test (creatinine-normalized [THC-COOH] ≥50 ng/mL).
4. Subjects must use inhalation (i.e., smoking, vaping) consistently as the primary route of cannabis administration. Additional use of edible cannabis is allowed.
5. Written informed consent to participate in the study.
6. Body mass index (BMI) between ≥18 and <35 kg/m2, inclusive, by Nomograph for BMI at screening.
7. Female subjects of childbearing potential, defined as having a menstrual cycle that is confirmed prior to enrollment, and who are heterosexually active and not surgically sterile or at least 2 years postmenopausal, must agree to use one of the following forms of contraception throughout the study and until 21 days after the last dose of study drug: abstinence, hormonal (oral, transdermal, implant, or injection), barrier (condom, diaphragm with spermicide), intrauterine device, or vasectomized partner (6 months minimum).
8. Male subjects are to refrain from donating sperm and heterosexually active male subjects must agree to the use of highly effective contraceptive methods (e.g., double barrier with at least condoms and spermicide) from screening through 90 days after the last dose of study drug, or their female partner must use a highly effective method of contraception as listed in inclusion criteria 7 from screening through 90 days after the last dose.
9. No clinically significant abnormal findings in the medical history, on physical examination, ECG, or clinical laboratory results (see Appendix B) during screening that could jeopardize the safety of the subject or impact the validity of the study.
10. Subjects must agree to return to the study site as required, be able to read English, and be willing to comply with all required study procedures.

Exclusion Criteria:

1. A history of clinically significant gastrointestinal, renal, hepatic, neurologic, hematologic, endocrine, oncologic, pulmonary, immunologic, psychiatric, or cardiovascular disease, or any other condition which, in the opinion of the principal investigator, would jeopardize the safety of the subject or impact the validity of the study results. For psychiatric disease, see more details below.
2. Subject has had significant traumatic injury, major surgery, or open biopsy within 30 days prior to the screening visit.
3. Presence or history within 12 months prior to screening of other substance use disorders according to DSM-5 criteria (as assessed by the MINI-5, psychiatric assessment, urine drug screen, breath analyzer, as appropriate) except for mild alcohol use disorder (as defined in DSM-5) or tobacco use disorder. Current use (within 30 days prior to screening) of opioid agonist or antagonist.
4. Subjects meeting DSM-5 criteria for schizophrenia, schizoaffective illness, or bipolar disorder. Subjects experiencing psychotic events which require psychiatric intervention or would interfere with study participation, apart from transient psychotic events due to substance abuse.
5. Subjects diagnosed with major depression and with a severity score of >17 based on HAM-D. Furthermore, subjects with other psychiatric disorders (excluding CUD) and with either a severity score at baseline of >4 based on CGI for other psychiatric disorders, or who have not been stable for at least the last 3 months prior to screening with either behavioral treatment or unchanged medication and dose. Subjects with a current psychiatric disorder treated with prohibited medications .
6. Subjects with a history of or current homicidal ideations or attempts.
7. Subjects with any suicidal behavior or answering 'yes' to question 4 or 5 on suicidal ideation within the past 2 years based on the Baseline/Screening version of the C-SSRS. Subjects with any suicidal behavior or answering 'yes' to question 4 or 5 on suicidal ideation longer than 2 years ago based on the Baseline/Screening version of the C-SSRS and who, in the opinion of the principal investigator, could be at risk of jeopardizing his/her own safety during the study
8. Subjects who use daily supplements of steroids (or food containing steroids), including pregnenolone, during the 4 weeks prior to the first screening visit. Topical use of steroids is allowed, and hormonal contraceptives are allowed if using a stable regimen throughout the study.
9. Subjects with frequent regular use of diet or supplements (e.g., St. John's Wort), food or grapefruit juice that may interfere with the activities of CYP P450.
10. Participation in a clinical trial within 1 month prior to the first dose of study drug, or 2 months if terminal half-life of the investigational drug is more than 120 hours.
11. Female subjects who are trying to conceive, are pregnant, are lactating or have a positive serum pregnancy test at screening or a positive urine pregnancy test at study visits, regardless of childbearing potential.
12. A positive urine drug screen for other drugs of abuse other than cannabinoids and/or a positive breath test for alcohol. One repeat alcohol breath test is allowed at a second screening visit or at the baseline visit.
13. Subjects with known allergy to corn or corn derivatives.
14. Legal status of the subject that in the opinion of the investigator would interfere with participation, e.g., risk of incarceration.
15. Subjects taking any of the medications or substances

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 333 (Actual)
Dates: Start 2022-05-06 (Actual); Primary Completion 2024-04-11 (Actual); Study Completion 2024-07-22 (Actual)

PRIMARY OUTCOMES:
Assessment of cannabis use | up to 16 weeks (end of study)
  Cannabis use will be assessed using self-reporting and monitored daily, prospectively by an EMA using a smartphone-based application
Assessment of cannabis use | up to 16 weeks (end of study)
  Cannabis use will be assessed using self-reporting and monitored daily, by using the TLFB procedure at each visit. The TLFB will be used to corroborate data obtained with EMA evaluation of cannabis use.

SECONDARY OUTCOMES:
Measures subject-rated intensity of withdrawal symptoms | up to 16 weeks (end of study)
  The 19-item version of the Cannabis Withdrawal Scale (CWS) that will be used measures subject-rated intensity of withdrawal symptoms as well as the amount of distress or impairment in functioning due to each symptom for the last 24 hours on a scale of 0 ("not at all") to 10 ("extremely"). The following statements describe how you have felt over the last 24 hours
Complete psychiatric diagnosis | up to 16 weeks (end of study)
  The MINI International Neuropsychiatric Interview (MINI-5) will be used in order to complete psychiatric diagnostic assessment to assess for CUD criteria in addition to other psychiatric disorders for eligibility.
Assesment of Quality of life | up to 16 weeks (end of study)
  the Patient-Reported Outcomes Measurement Information System-29 is a 29-item self-report measure to assess quality of life by assessing functioning and well-being in physical, mental, and social domains of health over the last 7 days.

OTHER OUTCOMES:
Assessment of Marijuana Craving | up to 16 weeks (end of study)
  The Marijuana Craving Questionnaire-Short Form (MCQ-12) is a 12-item self-report measures subjects' craving for marijuana on a Likert scale of 1-7 and yields total scores and factor scores in the areas of compulsivity, emotionality, expectancy, and purposefulness.
Assessment of Quality of sleep | up to 16 weeks (end of study)
  The Medical Outcome Study - Sleep Scale (MOS-SS) is a 12-item measure for characterizing the quality of sleep over the past 4 weeks.
Assessment of severity of nicotine dependence | up to 16 weeks (end of study)
  The Fagerstrom Test for Nicotine Dependence is a 6 item self-report questionnaire assessing severity of nicotine dependence
Assessment of desire to quit cannabis | up to 16 weeks (end of study)
  the Motivation to Quit Ladder is a single item change ladder from 1 to 10, where 1 is "no desire to quit" and higher numbers are greater desire to quit

CONTACTS AND LOCATIONS:
Overall Officials: Frances Levin, MD, Principal Investigator — Columbia University/NYSPI; Jennifer Wisdom, MD, Principal Investigator — CODA Inc, Research Department; Kevin Gray, MD, Principal Investigator — Addiction Sciences Division - Medical University of South Carolina; Jennifer Potter, MD, Principal Investigator — Department of Psychiatry and Behavioral Sciences - UT Health San Antonio.; Larissa Mooney, MD, Principal Investigator — Department of Psychiatry and Biobehavioral Sciences - UCLA; Rajita Sinha, MD, Principal Investigator — Addiction Program- Yale Stress Center; Richi Kakar, MD, Principal Investigator — Segal Trials; Paul Thielking, MD, Principal Investigator — CEDAR Salt Lake city; Olga Lapeyra, MD, Principal Investigator — Behavioral Clinical Research; Haig Goenjian, MD, Principal Investigator — CEnExel CNR; Matt Evans, MD, Principal Investigator — CEDAR Arizona
Locations (11):
- United States (11):
  - Cedar clinical research, Phoenix, Arizona
  - CenExel CNR, Garden Grove, California
  - UCLA Department of Psychiatry and Biobehavioral Sciences, Los Angeles, California
  - Yale Stress Center - Addiction Program, New Haven, Connecticut
  - Segal Trial, Lauderhill, Florida
  - Behavioral Clinical Research, Miami Lakes, Florida
  - The Substance Treatment and Research Service (S.T.A.R.S.) of Columbia University/NYSPI., New York, New York
  - CODA, Inc Research Department, Portland, Oregon
  - Addiction Sciences Division Department of Psychiatry and Behavioral Sciences Medical University of South Carolina, Charleston, South Carolina
  - Department of Psychiatry and Behavioral Sciences at UT Health San Antonio., San Antonio, Texas
  - Cedar Clinical Research, Draper, Utah

IPD SHARING:
Plan to Share IPD: No